CLINICAL TRIAL: NCT05053685
Title: Utility of Plasma and Urine Metanephrines in the Diagnosis of Phaeochromocytoma in Patients With Obstructive Sleep Apnoea
Brief Title: Metanephrines in Obstructive Sleep Apnoea
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OSA_Mets
Record Dates: First submitted 2021-09-12; First posted 2021-09-22 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-08

CONDITIONS: Pheochromocytoma; Obstructive Sleep Apnea; Catecholamine; Secretion
MeSH Terms: conditions — Pheochromocytoma; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obstructive Sleep Apnoea (OSA): Subjects with OSA
  Interventions: Diagnostic Test: Measurement of Urine and plasma metanephrines
- Elevated Urine Metanephrines: Subjects with elevated metanephrines
  Interventions: Diagnostic Test: Measurement of Urine and plasma metanephrines

INTERVENTIONS:
Diagnostic Test: Measurement of Urine and plasma metanephrines — Measurement of Urine and plasma metanephrines

SUMMARY:
Although most patients have essential (unexplained) hypertension, some patients have a treatable underlying condition. One such condition is phaeochromocytoma, a tumour that produces excessive stress hormones. Left undiagnosed, patients may develop a hypertensive crisis that can be fatal. Measurements of stress hormones (both 24-hour urine collection and morning blood tests) are highly sensitive for detecting these tumours. However, these stress hormones may also be elevated in obstructive sleep apnoea (OSA) which affects 1 in 5 adults.

The investigators hypothesize that in patients with OSA, blood tests will be better than 24-hr urine tests at ruling out a tumour. If this is confirmed, then OSA patients with suspected phaeochromocytoma could be investigated with a morning blood test instead of a traditional urine test, reducing unnecessary additional tests and patient anxiety.

In this single site study, the investigators plan to recruit 70 patients undergoing polysomnography. 24hr urine and bloods will be measured. Patients with elevated hormone levels will undergo imaging to rule out a tumour.

The primary outcome will be the accuracy of each test in ruling out a tumour. The secondary outcomes will be the relationship between stress hormone level and severity of OSA, which may help to explain the increased cardiovascular risk in patients with OSA, and the change in stress hormone level with treatment for OSA

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-70 years attending for a sleep study to evaluate for OSA

Exclusion Criteria:

* Medications that can cause changes in metanephrine levels
* Other factors that can cause changes in metanephrine levels
* Renal impairment (eGFR < 60ml/min)
* Other serious medical conditions

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending for sleep studies for evaluation of OSA
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Urine and plasma metanephrines | 1 year
  Measurement of 24 hours urine metanephrines
Urine and plasma metanephrines | 1 year
  Measurement of plasma metanephrines

SECONDARY OUTCOMES:
Relationship between metanephrine level and severity of OSA | 1 year
  comparison of metanephrine level and severity of OSA as dertermined by sleep study
Change in metanephrine levels with treatment for OSA | 1 year
  Change in plasma and urine metanephrine levels during treatment for OSA

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No